CLINICAL TRIAL: NCT02297672
Title: Partial Breast Irradiation Using Interstitial Permanent Palladium-103 Seed Implant
Acronym: PBSI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Juanita Crook, Radiation oncologist, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H14-02175
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Early Stage Breast Cancer
Keywords: breast cancer; brachytherapy; partial breast radiotherapy; palladium 103
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast seed implant (Experimental): Stranded palladium seed interstitial radioactive seed implant to seroma with margin with 3 dimensional ultrasound and CT guidance
  Interventions: Radiation: Stranded palladium seed interstitial implant; Device: 3 dimensional breast ultrasound; Device: Computerized tomography (CT)

INTERVENTIONS:
Radiation: Stranded palladium seed interstitial implant — Interstitial implantation of stranded palladium 103 seeds in seroma with a margin
Device: 3 dimensional breast ultrasound — guidance of placement of interstitial needles in breast
Device: Computerized tomography (CT) — Breast CT for planning and assessing interstitial implantation of radioactive seeds

SUMMARY:
Permanent Breast Seed Implant (PBSI) has been demonstrated to be a well accepted and well tolerated form of partial breast radiotherapy. This protocol aims to build on the initial experience and to further refine the technique and collect toxicity and cost data, especially in comparison to alternate forms of breast radiotherapy.

DETAILED DESCRIPTION:
25 women with low stage (pT1pN0) breast cancer, grade 1 or 2, will be accrued for adjuvant partial breast radiotherapy using PBSI and prospectively followed for 5 years. The primary aims is to evaluate implant quality according to recognized dosimetric parameters. Secondary aims include elaboration of approaches to different technical scenarios imposed by variation in seroma size, shape and location within the breast (expanding the technical manual to include recommended approaches to implants in different sectors of the breast and in different size breasts), incorporation of the use of live 3D ultrasound in the procedure (as opposed to current use of 2D US), assessment of patient acceptance and quality of life, physician assessment of cosmesis, assessment of toxicity, and recording of cost to the patient and health care system compared to alternate forms of breast radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent and signature of approved consent form.

  * Age greater than 55 years and postmenopausal.
  * Life expectancy of at least ten years
  * Stage 0 or I breast cancer. Tumour size < 2 cm.
  * Invasive cancer must be pathologic grade 1 or 2
  * Histology must be either Ductal Carcinoma In Situ or invasive ductal adenocarcinoma of the breast.
  * Tumour removed by lumpectomy with clear margins (DCIS and invasive).
  * Unifocal disease
  * For invasive breast cancer, axillary staging by either sentinel node biopsy or axillary dissection (minimum of 6 axillary nodes). Not required for DCIS.
  * Brachytherapy generally should be performed within 16 weeks of the last surgery (lumpectomy, re-excision of margins, or axillary staging procedure). If > 16 weeks, will be assessed on case-by-case basis, based on seroma visibility and the presence of surgical clips in the tumour bed.
  * Tumour must be Estrogen Receptor positive.
  * The lumpectomy cavity (seroma) must be clearly delineated by ultrasound and CT and should be < 3 cm diameter (equivalent sphere) resulting in a maximum of 125 cc planning target volume (PTV).
  * Breast seed implant must be considered technically deliverable by interstitial brachytherapy by the attending radiation oncologist and must be a minimum 2-plane implant.
  * If prior non-breast malignancies, must have been disease-free for 5 or more years. Time limit waived for carcinoma in-situ of the cervix or colon, melanoma in-situ, and basal or squamous cell carcinoma of the skin.

Exclusion Criteria:

* Stage T2 or higher breast cancer

  * Histologically positive axillary nodes.
  * High grade (grade 3) invasive ductal carcinoma
  * Extensive DCIS
  * Lymphatic or Vascular Invasion positive
  * Significant persistent post surgical complications
  * Palpable or radiographically suspicious ipsilateral or contralateral axillary, or regional nodes, unless histologically confirmed negative.
  * Suspicious microcalcifications, densities, or palpable abnormalities in the ipsilateral or contralateral breast unless confirmed benign.
  * Proven multi-centric carcinoma (invasive cancer or DCIS)
  * Paget's disease of the nipple.
  * Synchronous bilateral invasive or non-invasive breast cancer.
  * History of previous ipsilateral invasive breast cancer or DCIS.
  * Surgical margins that are positive or cannot be microscopically assessed.
  * Clear delineation of the target lumpectomy cavity not possible.
  * Breast implants.
  * Prior ipsilateral breast or thoracic radiotherapy.
  * Known genetic mutation in Breast Cancer Associated (BRCA 1 or 2)
  * Collagen vascular disease,

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Implant quality | Day 0
  Post implant CT evaluation to report dosimetric parameters including the minimum dose in Gray to 90% of the target volume (D90) and the percentage of the target volume (seroma, seroma with 5 mm margin, seroma with 10 mm margin) receiving 100% of the prescribed dose (V100).

SECONDARY OUTCOMES:
Eligibility for implant based on seroma size and location within breast | Day 0
  US and CT evaluation to record the range of seroma volumes and quadrant location in the breast acceptable for implantation
Feasibility of 3D US for procedure guidance | Day 0
  Post implant CT evaluation describing dosimetric parameters (D90 and V100 as above in Outcome 1) with the use of 3D ultrasound and with 2D ultrasound
Cosmesis | 5 years
  Physician assessed using the questionnaire from the Radiation Therapy Oncology Group (RTOG) and National Surgical Adjuvant Breast Project (NSABP)
Acute and Late Toxicity of breast brachytherapy | 5 years
  Physician assessed using the Common Terminology Criteria for Adverse Events (CTCAE V4) form
Patient Assessed Quality of life using the NSABP/RTOG breast Cancer Quality of Life questionnaire | 3 years
  Patient assessed using the RTOG/NSABP Breast Cancer Quality of Life Assessment form
Dose to Organs at risk | Day 0
  Post implant CT assessment describing calculated doses to lung, ribs and heart described as the highest dose to 1 cc of the specific organ tissue and skin dose recorded as an area 1 cm by 1 cm by 2 mm thick (1cmx1cmx0.2cm)
Cost | 5 years
  Cost to health care system (Canadian dollars) and patient (expenses and lost wages in Canadian dollars)

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Crook, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BCCA Center for the Southern Interior, Kelowna, British Columbia, Canada

REFERENCES:
- [Result] Pignol JP, Keller B, Rakovitch E, Sankreacha R, Easton H, Que W. First report of a permanent breast 103Pd seed implant as adjuvant radiation treatment for early-stage breast cancer. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):176-81. doi: 10.1016/j.ijrobp.2005.06.031. Epub 2005 Sep 22. PMID 16182464
- [Result] Keller BM, Ravi A, Sankreacha R, Pignol JP. Permanent breast seed implant dosimetry quality assurance. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):84-92. doi: 10.1016/j.ijrobp.2011.05.030. Epub 2011 Oct 20. PMID 22019237
- [Result] Olivotto IA, Whelan TJ, Parpia S, Kim DH, Berrang T, Truong PT, Kong I, Cochrane B, Nichol A, Roy I, Germain I, Akra M, Reed M, Fyles A, Trotter T, Perera F, Beckham W, Levine MN, Julian JA. Interim cosmetic and toxicity results from RAPID: a randomized trial of accelerated partial breast irradiation using three-dimensional conformal external beam radiation therapy. J Clin Oncol. 2013 Nov 10;31(32):4038-45. doi: 10.1200/JCO.2013.50.5511. Epub 2013 Jul 8. PMID 23835717